CLINICAL TRIAL: NCT07255482
Title: Mortality Benefit of Ultrasound for Incidental Thyroid Nodules Identified With PET Imaging: A Non-Inferiority Emulated Target Trial
Brief Title: Mortality Benefit of Ultrasound for Thyroid Nodules Identified With PET Imaging: Non-Inferiority Emulated Target Trial
Status: Active, not recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jeffrey P Guenette, Associate Professor of Radiology, Brigham and Women's Hospital
Other Study IDs: 2024P002073-1; R18HS029839 (AHRQ)
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Thyroid Nodule (Benign); Thyroid Nodule (Diagnosis); Thyroid Cancer
MeSH Terms: conditions — Thyroid Nodule; Disease; Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with thyroid nodule on PET
  Interventions: Diagnostic Test: Thyroid Ultrasound

INTERVENTIONS:
Diagnostic Test: Thyroid Ultrasound — Thyroid ultrasound performed within 3 months of PET to characterize a thyroid nodule identified on the PET

SUMMARY:
The investigators hypothesize that all-cause mortality in patients with an incidental thyroid nodule on PET-CT who did not have thyroid ultrasound (the exposure) within 3 months of the PET-CT is non-inferior within a 5% margin to those who have thyroid ultrasound at 7-years. That is, among patients with an incidental thyroid nodule on PET-CT, mortality is no more than 5% larger (in absolute difference) for those who do not have thyroid ultrasound compared to those who do. The investigators will also report mortality differences at landmark timeframes of 1-year, 3-years, 5-years, and 10-years. To estimate group differences in mortality, the investigators will conduct a non-inferiority emulated target trial utilizing clone-censor weighting to address potential immortal time bias introduced by the 3-month grace period. The investigators will adjust for demographic, potential confounder, and mortality risk adjustor factors. The investigators will stratify analyses based on baseline disease severity (estimated 5-year relative survival risk) and disease status (progression, lymph node involvement, other sites of metastases). All subjects will be accrued from the Mass General Brigham healthcare system, which includes two academic medical centers, a specialty head and neck hospital, and multiple community hospitals and numerous community clinics.

DETAILED DESCRIPTION:
Study Hypothesis: The investigators hypothesize that all-cause mortality in patients with an incidental thyroid nodule on PET-CT who did not have thyroid ultrasound within 3 months is no worse than 5% lower than those who did have ultrasound.

Outcome Measures:

Primary Outcome: All-cause mortality. Secondary Outcomes: Numbers of thyroid cancer diagnoses, thyroid ultrasounds, thyroid biopsies, and thyroid surgeries Exploratory Outcomes: Types of thyroid cancer diagnoses

Study Population: All patients age 18-years and older with incidental thyroid nodule on PET-CT performed between 1/1/2015 and 12/31/2021.

Sites/Facilities: Mass General Brigham healthcare system including Massachusetts General Hospital, Brigham and Women's Hospital, Mass Eye and Ear, and associated community sites.

Exposure: Thyroid ultrasound evaluation within 3-months of PET-CT.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=18
2. Thyroid nodule on PET-CT performed 1/1/2015 to 12/31/2021
3. At least one clinical note in the EHR from the 36-month window prior to the PET

Exclusion Criteria:

1. Thyroid ultrasound listed in the medical record in the prior 3 years
2. Documented history of prior thyroid cancer diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had a PET-CT at Mass General Brigham 1/1/2015 to 12/31/2021
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
All-Cause Mortality | 7 Years

SECONDARY OUTCOMES:
Number of Thyroid Cancer Diagnoses | 7 Years
Number of Thyroid Ultrasound Examinations | 7 Years
Number of Thyroid Biopsies | 7 Years
Number of Thyroid Surgeries | 7 Years

OTHER OUTCOMES:
Types of Thyroid Cancers | 7 Years
  Exploratory

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
All deidentified data used in the study analysis.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Study protocol with study analysis plan submitted at time of clinicaltrials.gov registration. IPD and analytic code will be shared upon manuscript publication.
Access Criteria: General public via the Harvard Dataverse repository.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-20): https://cdn.clinicaltrials.gov/large-docs/82/NCT07255482/Prot_SAP_000.pdf